CLINICAL TRIAL: NCT04792255
Title: Investigation of Dose Management Capabilities of Digital Variance Angiography: Contrast Media Dose Reduction in Patients Undergoing Carotid Artery Stenting - a Prospective Randomized Clinical Trial
Brief Title: Digital Variance Angiography for Contrast Media Dose Reduction in Carotid Artery Stenting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kinepict Health Ltd. (Network)
Collaborators: Semmelweis University (Other); Bács-Kiskun County Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Kinepict-009
Record Dates: First submitted 2021-02-23; First posted 2021-03-10 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-07

CONDITIONS: Carotid Artery Diseases
Keywords: Radiocontrast media reduction; X-ray angiography; Digital Variance Angiography; Digital Subtraction Angiography; carotid artery stenting; Kinepict
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Vascular Access Devices

STUDY DESIGN:
Intervention Model Description: Enrolled participants will undergo carotid artery stenting with different image acquisition protocol of the pre-and postinterventional angiographies from anteroposterior and lateral views, and intraoperative angiographies with C-arm angulations based on the operator's decision. In the active comparator group, a standard contrast media dose and DSA images will be used for diagnosis whereas in the experimental group a reduced contrast media dose will be applied (50% decrease compared to the standard DSA protocol) and the operator will use DVA images for the diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Reduced contrast media dose group (Experimental): Reduced contrast media protocol: extracranial carotid artery intervention (2-4 fps according to the institutional protocol).
  Contrast administration with an automatic contrast injector: angiographic image acquisitions will be performed with 6 ml of 50% contrast media (3 ml iodined contrast media, 3 ml physiologic saline) with a 3 ml/s flow rate.
  DSA and DVA images will be calculated; DVA images will be used for diagnosis and interventions.
  Interventions: Procedure: Carotid artery stenting with reduced contrast media protocol; Diagnostic Test: Carotid Duplex Ultrasound
- Group B: Standard contrast media dose group (Active Comparator): Standard contrast media protocol: extracranial carotid artery intervention (2-4 fps according to the institutional protocol).
  Contrast administration with an automatic contrast injector: angiographic image acquisitions will be performed with 6 ml iodined contrast media with a 3 ml/s flow rate.
  DSA and DVA images will be calculated; DSA images will be used for diagnosis and interventions.
  Interventions: Procedure: Carotid artery stenting with standard contrast media protocol; Diagnostic Test: Carotid Duplex Ultrasound

INTERVENTIONS:
Procedure: Carotid artery stenting with standard contrast media protocol — Radial, brachial or femoral arterial access is gained by using the Seldinger technique. The common carotid artery (CCA) is catheterized. Selective angiography is performed from the anteroposterior and lateral view without magnification. Initial angiograms are performed with standard contrast media protocol in anteroposterior and lateral views without magnification with the sheath placed in the common carotid artery. The carotid arterial lesion is crossed and an embolic protection device is deployed in the internal carotid artery. Carotid artery stenting is performed in a standard fashion. Post-stenting angiographies are obtained with the standard contrast media protocol in anteroposterior and lateral views without magnification with the sheath placed in the CCA. Pre- and post-stenting angiographies are performed with the same sheath position. DSA and DVA images will be calculated on a commercially available image processing workstation and the Kinepict Medical Imaging Tool.
  Other Names: Arterial access; Preinterventional selective carotid artery angiography; Carotid artery stenting; Postinterventional selective carotid artery angiography
  Arms: Group B: Standard contrast media dose group
Procedure: Carotid artery stenting with reduced contrast media protocol — Radial, brachial or femoral arterial access is gained by using the Seldinger technique. The common carotid artery (CCA) is catheterized. Selective angiography is performed from the anteroposterior and lateral view without magnification. Initial angiograms are performed with the reduced contrast media protocol in anteroposterior and lateral views without magnification with the sheath placed in the common carotid artery. The carotid arterial lesion is crossed and an embolic protection device is deployed in the internal carotid artery. Carotid artery stenting is performed in a standard fashion. Post-stenting angiographies are obtained with the reduced contrast media protocol in anteroposterior and lateral views without magnification with the sheath placed in the CCA. Pre- and post-stenting angiographies are performed with the same sheath position. DSA and DVA images will be calculated on a commercially available image processing workstation and the Kinepict Medical Imaging Tool.
  Other Names: Arterial access; Preinterventional selective carotid artery angiography; Carotid artery stenting; Postinterventional selective carotid artery angiography
  Arms: Group A: Reduced contrast media dose group
Diagnostic Test: Carotid Duplex Ultrasound — Pre- and postinterventional assessment of the treated internal carotid artery.

SUMMARY:
Digital Variance Angiography (DVA) is a new tool in medical imaging with a proven image quality reserve (1, 2).

Previous studies have demonstrated the quality reserve of DVA in angiographic studies (1, 2), which allowed us to reduce contrast media use by 50% in carotid artery angiographic studies without affecting the image quality (3).

CAS is an alternative treatment option for carotid artery revascularization in selected patient groups. Similar to most of the minimally invasive endovascular interventions, CAS also carries the risk of contrast-induced acute kidney injury, which is considered to be an independent predictor of 30-day major adverse events (4).

The aim of this study is to apply DVA in patients undergoing carotid artery stenting (CAS) and utilize this technique to reduce contrast dose during the interventions, without affecting the intraprocedural radiation dose and the clinical outcome of the procedures. Investigators believe that the reduction in contrast media use and the associated image quality with the technique of DVA imaging can be incorporated into the everyday clinical practice, and will play an important role in improving the rate of contrast-induced acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y
* Carotid stenosis defined as:

Stenosis ≥70% by computer tomography angiography (NASCET criteria); OR by duplex-ultrasound with ≥70% stenosis defined by a peak systolic velocity of at least 230 cm/s

* Carotid stenosis is treatable with CAS

Exclusion Criteria:

* History of stroke or TIA ipsilateral to the stenosis within 30 days of randomization
* Acute myocardial infarction
* Severe chronic kidney disease: GFR>30ml/min/m2
* Severe heart failure: NYHA IV
* Severe liver failure: Child-Pugh 3
* Iodine contrast allergy
* Coagulopathy
* Hematological bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
DSA-related contrast media use | During the procedure
  Volume of the iodinated contrast agent used for enhancing the image quality (mL)
Total procedural contrast media use | During the procedure
  Volume of the iodinated contrast agent used for enhancing the image quality (mL)
Image quality, graded by independent observers | through study completion, an average of 1 year
  Observations based on a 5-level Likert scale (1-poor image quality, 3-medium image quality, 5-outstanding image quality)

SECONDARY OUTCOMES:
Total procedural dose area product | During the procedure
  Indicator of a patient's irradiation dosage (microGy*cm2 or Gy*cm2)
DSA-related dose area product | During the procedure
  Indicator of a patient's irradiation dosage (microGy*cm2 or Gy*cm2)
Total procedural time | During the procedure
  Duration of the whole procedure, from arterial access till the removal of every tool (min)
Number of protocol changes during DVA usage | During the procedure
  Number of occasions when the reduced contrast media protocol has to be switched back to conventional protocol because of the unsuitable image quality
Residual stenosis | During the procedure
  The difference between the normal reference segment diameter and the minimum lumen diameter of the treated lesion after CAS (%)
Focal neurological symptoms | During the procedure and up to 1 day
  Focal neurological symptoms ipsilateral to the treated carotid artery during the postprocedural observation period
Preoperative and postoperative ipsilateral carotid artery flow by doppler ultrasound | Preoperatively and 1 day after the procedure
  Peak-systolic and end-diastolic velocities (cm/sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Heart and Vascular Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gyano M, Gog I, Orias VI, Ruzsa Z, Nemes B, Csobay-Novak C, Olah Z, Nagy Z, Merkely B, Szigeti K, Osvath S, Sotonyi P. Kinetic Imaging in Lower Extremity Arteriography: Comparison to Digital Subtraction Angiography. Radiology. 2019 Jan;290(1):246-253. doi: 10.1148/radiol.2018172927. Epub 2018 Oct 16. PMID 30325284
- [Background] Orias VI, Gyano M, Gog I, Szollosi D, Veres DS, Nagy Z, Csobay-Novak C, Zoltan O, Kiss JP, Osvath S, Szigeti K, Zoltan R, Sotonyi P. Digital Variance Angiography as a Paradigm Shift in Carbon Dioxide Angiography. Invest Radiol. 2019 Jul;54(7):428-436. doi: 10.1097/RLI.0000000000000555. PMID 30829769
- [Background] Orias VI, Szollosi D, Gyano M, Veres DS, Nardai S, Csobay-Novak C, Nemes B, Kiss JP, Szigeti K, Osvath S, Sotonyi P, Ruzsa Z. Initial evidence of a 50% reduction of contrast media using digital variance angiography in endovascular carotid interventions. Eur J Radiol Open. 2020 Nov 17;7:100288. doi: 10.1016/j.ejro.2020.100288. eCollection 2020. PMID 33294499
- [Background] Paraskevas KI, Mikhailidis DP. Contrast-Induced Acute Kidney Injury in Patients Undergoing Carotid Artery Stenting: An Underestimated Issue. Angiology. 2017 Oct;68(9):752-756. doi: 10.1177/0003319716668934. Epub 2016 Sep 19. PMID 27645233